CLINICAL TRIAL: NCT01360190
Title: Neurophysiologic Monitoring of Antidepressant Treatment
Acronym: Lilly
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Andrew F. Leuchter, MD, UCLA Laboratory of Brain, Behavior, and Pharmacology
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 94-08-273-13
Record Dates: First submitted 2011-05-23; First posted 2011-05-25 (Estimated); Last update posted 2011-05-25 (Estimated); Status verified 2011-05

CONDITIONS: Major Depressive Disorder
Keywords: MDD; major depressive disorder; QEEG; electroencephalograph; fluoxtine; placebo
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Fluoxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- fluoxetine (Active Comparator)
  Interventions: Drug: fluoxetine
- placebo (Placebo Comparator)
  Interventions: Drug: fluoxetine

INTERVENTIONS:
Drug: fluoxetine — fluoxetine 20 mg. daily

SUMMARY:
The overall goal of this proposal is to study quantitative electroencephalography (QEEG ) as a method for the detection of antidepressant treatment response. The investigators have developed a QEEG algorithm called "cordance" that appears to provide much the same information about brain function as PET or SPECT scanning, and has shown patterns of brain function that appear to be indicative of depression. Of greatest interest is that these patterns appear to normalize in response to antidepressant treatment.

DETAILED DESCRIPTION:
Background and Significance/Preliminary Studies:

A. Cordance. There is considerable evidence indicating that abnormal slow-wave activity in the EEG is caused by partial cortical deafferentation. Despite this fact, no clinically relevant measure of deafferentation has been available. The investigators sought to develop such a measure by examining young and old subjects with white-matter lesions that presumably undercut the cerebral cortex, as well as subjects with several different types of brain disease who had undergone SPECT scanning. The investigators discovered an indicator termed discordance, that is characteristic of cortex undercut by white-matter lesions, or that is hypoperfused for any reason. The investigators also discovered an indicator the investigators termed concordance , which is characteristic of cortex that has normal perfusion.

This overall technique for the non-invasive assessment of afferent function, cerebral perfusion, and metabolism the investigators call cordance mapping, which is the subject of a United States patent. A detailed explanation of the formulae used to calculate cordance is provided in the manuscripts referenced above. The first of these two manuscripts contains illustrative examples where discordance was useful in detection of white-matter lesions or degenerative disease. The second manuscript shows a quantitative analysis of cordance and HMPAO-SPECT data from 27 patients with a variety of conditions, and demonstrates that cordance is superior to conventional EEG measures in its correlations with relative perfusion. Like SPECT, cordance measurements vary according to the patients' state, but has high test-retest reliability for detecting brain lesions.

B. Differential diagnosis of depression. One promising application of cordance is to the differential diagnosis of psychiatric illness. A "normal" cordance pattern is one of posterior dominant concordance with cordance values near zero in the frontal regions. The investigators have reported a "classic" cordance pattern for subjects with Alzheimer's disease (DAT), in which there is parietal discordance (in the beta or theta bands) in conjunction with alpha concordance that has shifted from the occipital to the central head regions. This finding is consistent with the pattern seen commonly on PET and SPECT, in which there is parietal hypoperfusion or hypometabolism with preserved metabolism over the central head regions (the motor strip), which is known to be less affected by Alzheimer's changes.

In evaluating treatment results, the investigators will need to determine what effect medication status has upon QEEG measures. Although results thus far suggest that there is little significant effect , the investigators will carefully examine the effects of antidepressant and antianxiety medications further

METHODS:

The investigators plan to examine cordance in 26 subjects undergoing antidepressant treatment, and to use this neurophysiologic method to assess the response to treatment in depressed patients. The project has the following three specific aims: 1) to identify physiologic indices of fluoxetine treatment response using quantitative EEG; 2) to detect how early in the course of fluoxetine treatment response this response may be detected; 3) to determine if QEEG measures of response distinguish subjects who are not responding to treatment from those who are responding.

The study will tests the hypothesis that those subjects receiving active treatment who show clinical improvement will demonstrate normalization of cordance maps. Conversely, the investigators hypothesize that those subjects who either do not show improvement, or who have some improvement on placebo, will not show normalization of cordance.

The investigators will examine these hypotheses with a four-step plan. Specifically, the investigators will recruit 26 patients with major depression and perform baseline assessments of the severity of depressive symptoms, as well as QEEG studies. Second, the investigators will enroll these patients in an eight-week, double-blind placebo-controlled study in which they will receive either fluoxetine 20 mg. daily or placebo. Third, the investigators will follow subjects with ratings of mood and serial QEEG studies to determine if there is an association between resolution of depressive symptoms and QEEG cordance changes. Fourth, the investigators will enroll subjects in open-label treatment at the end of the eight weeks and examine cordance in those who previously received placebo and, where appropriate, in those receiving fluoxetine 40 mg. daily.

ELIGIBILITY:
Inclusion Criteria:

* All subjects will meet DSM-IV criteria for major depression based upon the Structured Clinical Interview for DSM-IV - Patient Version (SCID-P) (First et al., 1994). All research personnel have undergone SCID-P training, and soon will extend this training to the DSM-IV version.
* Subjects also will have a score on the 17-item Hamilton Depression Rating Scale of > 18 (with item #1 > 2).
* All subjects will be under the care of a clinician not affiliated with the study at the time of entry into the study, and through the course of the study.

Exclusion Criteria:

* Subjects will have no serious medical illness.
* We will exclude patients also meeting criteria for the following groups of axis I diagnoses: delirium or dementia, substance-related disorders, schizophrenia or other psychotic disorders, or eating disorders.
* In addition, patients meeting criteria for cluster A or B axis II diagnoses will be excluded.
* Subjects with a history of current or past active suicidal ideation, or suicide attempts will be excluded, as will patients who previously have failed to respond to an adequate clinical trial of fluoxetine, or have failed to tolerate the medication.
* Subjects who have had suboptimal trials, however, may still be considered for the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 1994-08; Primary Completion 1996-08 (Actual); Study Completion 1996-08 (Actual)

PRIMARY OUTCOMES:
Change in Hamilton Rating Scale For Depression Score | baseline, end of placebo-lead-in; and 48 hours, 1 week, 2 weeks, 4 weeks, and 8 weeks after randomized treatment
  We will determine which subjects demonstrate improvement on the primary outcome measure (Ham-D) obtained the day of the EEG, and enter these as categorical variables (improved/not improved).

CONTACTS AND LOCATIONS:
Overall Officials: Andrew F Leuchter, Principal Investigator — University of California, Los Angeles